CLINICAL TRIAL: NCT02784600
Title: Rotation MEdical BioindUctive ImpLant Database (REBUILD) Registry
Brief Title: Rotation Medical Bioinductive Implant Database Registry
Acronym: REBUILD
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 3679-01
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Rotator Cuff Tear
Keywords: Partial-thickness; Full-thickness
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Partial or full-thickness rotator cuff tear: Rotation Medical bioinductive implant
  Interventions: Device: Bioinductive implant

INTERVENTIONS:
Device: Bioinductive implant
  Other Names: Rotation Medical Rotator Cuff System™

SUMMARY:
The purpose of this clinical registry is to prospectively collect and compare preoperative and postoperative patient-reported data using validated shoulder-specific and health-related quality of life (QoL) instruments during real-world use of the Rotation Medical bioinductive implant to treat rotator cuff tears.

ELIGIBILITY:
Inclusion Criteria:

1. At least 21 years of age.
2. Able and willing to provide voluntary consent to Registry participation.
3. Able to read, speak, and understand the English language.

Exclusion Criteria:

1. Hypersensitive to bovine-derived materials.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical registry will be a prospective, multi-center registry conducted under a common protocol where all subjects will undergo treatment with the Rotation Medical bioinductive implant.
Sampling Method: Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Shoulder pain | 1 year
  Change between baseline and post-operative shoulder pain over time using a Visual Analog Scale (VAS).
American Shoulder and Elbow Surgeons Standardized Form for the Assessment of the Shoulder (ASES) | 1 year
  Change between baseline and post-operative ASES shoulder score over time.
Single Assessment Numeric Evaluation (SANE) Score | 1 year
  Change between baseline and post-operative SANE score over time.
Veterans RAND 12 Item Health Survey (VR-12) | 1 year
  Change between baseline and post-operative VR-12 score over time.
Western Ontario Rotator Cuff Index (WORC) | 1 Year
  Change between baseline and post-operative WORC score over time.

SECONDARY OUTCOMES:
Safety assessed by number of Adverse Events and Serious Adverse Events. | 1 Year
  Safety will be evaluated by reporting any Adverse Events that occur over the duration of the study and calculating the overall occurrence rate of Adverse Events and Serious Adverse Events
Recovery by cumulative number of days shoulder is in a sling | 1 Year
Recovery by cumulative time in days between discharge and return to work. | 1 Year
Recovery by cumulative time between discharge and return to driving | 1 Year
Recovery by cumulative time days between discharge and return to overhead-throwing and non-overhead throwing sports | 1 Year
  Overhead-throwing sports overhead-throwing (e.g., baseball, football or exercise where arm extends above head) and non-overhead-throwing (e.g., running, bowling or exercise where arm DOES NOT extend above head) sports.
Recovery by cumulative number physical therapy (PT) visits to rehabilitate the index shoulder. | 1 Year
Recovery by cumulative number of days of narcotic medication use to manage post-operative shoulder pain. | 1 Year
Recovery by cumulative number corticosteroid injections used to manage post-operative shoulder pain. | 1 Year
Revision Surgery | 1 Year
  Number of participants with a revision surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Louis McIntyre, MD, Principal Investigator — Phelps Medical Associates; Rachael Winter, Study Chair — Smith & Nephew, Inc.
Locations (19):
- United States (19):
  - Orthopaedic Specialty Institute, Orange, California
  - Glenwood Orthopaedic Center, Glenwood Springs, Colorado
  - Andrews Research & Education Foundation, Gulf Breeze, Florida
  - Andrews Sports Medicine & Orthopaedic Center, Gulf Breeze, Florida
  - Jacksonville Orthopaedic Institute, Jacksonville, Florida
  - Schofield, Hand, & Bright Orthopaedics, Sarasota, Florida
  - Harbin Clinic Orthopaedics & Sports Medicine Rome, Rome, Georgia
  - OrthoIllinois, LTD, Rockford, Illinois
  - Norton Orthopaedic & Sports, Louisville, Kentucky
  - Orthopaedic Surgical Associates, North Chelmsford, Massachusetts
  - Advanced Orthopedics of Detroit, PC, Saint Clair Shores, Michigan
  - Atlantic Orthopaedics & Sports Medicine, Portsmouth, New Hampshire
  - Lourdes Medical Associates (LMA) Professional, Burlington, New Jersey
  - Stony Brook Orthopaedics, Setauket, New York
  - Westchester Medical Pavilion, White Plains, New York
  - Hand and Microsurgery Associates, Columbus, Ohio
  - Central Texas Sports Medicine & Orthopaedics, PA, Bryan, Texas
  - Bone & Joint Clinic of Houston, Houston, Texas
  - Plano Orthopedic Sports Medicine & Spine Center, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McIntyre LF, Bishai SK, Brown PB 3rd, Bushnell BD, Trenhaile SW. Patient-Reported Outcomes After Use of a Bioabsorbable Collagen Implant to Treat Partial and Full-Thickness Rotator Cuff Tears. Arthroscopy. 2019 Aug;35(8):2262-2271. doi: 10.1016/j.arthro.2019.02.019. Epub 2019 Jul 23. PMID 31350082